CLINICAL TRIAL: NCT05648526
Title: Neuroprotective Effects of ACTH4-10PRO8-GLY9-PRO10 on The Ketamine-Induced Neurotoxicity In Neonatal Rats: Increased BDNF Expression And BDNF Serum Concentrations
Brief Title: Neuroprotective Effects of ACTH4-10PRO8-GLY9-PRO10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Raka Jati Prasetya, Doctor, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intervention
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Ketamine-Induced Neurotoxicity
Keywords: ACTH4-10Pro8-Gly9-Pro10; BDNF; ketamine-induced neurotoxicity; apoptosis
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTH4-10PRO8-GLY9-PRO10 (Experimental): The compound ACTH4-10Pro8-Gly9-Pro10 is a synthetic analog molecule of a short fragment of adrenocorticotropic hormone (ACTH). It is free from hormonal effects and has neuromodulatory effects.
  Interventions: Drug: ACTH4-10Pro8-Gly9-Pro10
- ketamine 40 mg/kg BW subcutaneously (Active Comparator): ketamine results in impaired brain function associated with neuroapoptosis injury in the immature brain.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: ACTH4-10Pro8-Gly9-Pro10 — ACTH4-10Pro8-Gly9-Pro10 also has neuromodulator characteristics to function as a neuroprotector in inhibiting the apoptotic process. Modulation by ACTH4-10Pro8-Gly9-Pro10 will increase the levels of BDNF thereby inhibiting the process of apoptosis
  Arms: ACTH4-10PRO8-GLY9-PRO10
Drug: Ketamine — negative-positive control (ketamine 40 mg/kg BW subcutaneously)
  Arms: ketamine 40 mg/kg BW subcutaneously

SUMMARY:
The compound ACTH4-10Pro8-Gly9-Pro10 is a synthetic analog molecule of an adrenocorticotropic hormone (ACTH) short fragment. That is free from hormonal effects and has neuromodulatory effects. We investigate the neuroprotective effects of ACTH4-10Pro8-Gly9-Pro10 can lessen neurotoxicity against ketamine in neonatal rats by looking at BDNF expression in the cortex and hippocampus tissue as well as BDNF blood levels.

DETAILED DESCRIPTION:
The compound ACTH4-10Pro8-Gly9-Pro10 is a synthetic analog molecule of a short fragment of adrenocorticotropic hormone (ACTH). It is free from hormonal effects and has neuromodulatory effects. The immune-modulating and neurotrophic activity of the drug were shown to balance the state of anti-inflammatory and trophic factors (IL-IO, TNF-a, TGF-Pl, BDNF, NGF) over proinflammatory factors (IL-Ip, IL-8, CRP, LE) to increase the anti-apoptotic defense (Bcl-2 elevation), as well as to reduce the peroxidation process (increased SOD activity).

ACTH4-10Pro8-Gly9-Pro10 also has neuromodulator characteristics to function as a neuroprotector in inhibiting the apoptotic process. Modulation by ACTH4-10Pro8-Gly9-Pro10 will increase the levels of BDNF thereby inhibiting the process of apoptosis. Based on research by Gusev and Skvortsova, ischemic stroke patients who were given ACTH4-10Pro8-Gly9-Pro10 showed increased levels of BDNF, decreased mortality, and reduced length of stay. Based on the description above, the researcher was interested in analyzing the effect of the administration of ACTH4-10Pro8-Gly9-Pro10 on ketamine neurotoxicity in neonatal rats by assessing the level of BDNF.

ELIGIBILITY:
Inclusion Criteria:

* Rattus norvegicus rats
* Male, seven days old, weighing 15-20 grams
* Spraque-Dawley strain, obtained from the Experimental Animal Care Unit

Exclusion Criteria:

* Animals that behave aggressively in observation by attacking other groups

Ages: 7 Days to 7 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
BDNF Expression | On 6 hours after the study drug dose
  a protein that, in humans, is encoded by the BDNF gene
BDNF Serum Concentrations | On 6 hours after the study drug dose
  a protein that, in humans, is encoded by the BDNF gene

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ing C, DiMaggio C, Whitehouse A, Hegarty MK, Brady J, von Ungern-Sternberg BS, Davidson A, Wood AJ, Li G, Sun LS. Long-term differences in language and cognitive function after childhood exposure to anesthesia. Pediatrics. 2012 Sep;130(3):e476-85. doi: 10.1542/peds.2011-3822. Epub 2012 Aug 20. PMID 22908104
- [Result] Flick RP, Katusic SK, Colligan RC, Wilder RT, Voigt RG, Olson MD, Sprung J, Weaver AL, Schroeder DR, Warner DO. Cognitive and behavioral outcomes after early exposure to anesthesia and surgery. Pediatrics. 2011 Nov;128(5):e1053-61. doi: 10.1542/peds.2011-0351. Epub 2011 Oct 3. PMID 21969289